CLINICAL TRIAL: NCT03937466
Title: Reducing the Experience of Menopausal Symptoms Through Temperature (REST)
Brief Title: Reducing the Experience of Menopausal Symptoms Through Temperature
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00057388
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Hot Flashes; Menopause
Keywords: hot flashes; menopause; cooling mattress pad
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Intervention Model Description: 24 peri or postmenopausal women aged 45-60 experiencing at least 4 hot flashes/night sweats/day will use a cooling mattress pad nightly for approximately 8 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental Cooling Mattress Pad (Experimental): Subjects will use a cooling mattress pad nightly for approximately 8 weeks
  Interventions: Device: Cooling mattress pad

INTERVENTIONS:
Device: Cooling mattress pad — The cooling mattress pad is a commercially available pad designed to be placed between the top of a mattress and bed sheets. It allows for precise temperature regulation in one's bed.

SUMMARY:
The purposes of this study are to obtain preliminary evidence on the efficacy of a cooling mattress pad in reducing subjective hot flashes for peri and postmenopausal women experiencing menopausal hot flashes, and to obtain preliminary evidence on the efficacy of a cooling mattress pad for improving sleep for peri and postmenopausal women experiencing menopausal hot flashes.

DETAILED DESCRIPTION:
Women will be recruited from the community through flyers. They will call into a study phone line at which time they will be screened for their initial eligibility using a telephone screener. Women who are eligible and willing to participate, will either come to the Research Center in Winston-Salem to be consented and complete baseline questionnaires or complete these by mail or email. After two weeks, women will mail back their diaries and continue to record their daily hot flashes until they are notified by study staff of their eligibility, within a week of receiving the diary. If they qualify, a cooling mattress pad will be provided by study staff to be used for the duration of the intervention phase for approximately 8 weeks. The study staff will determine the efficacy of the cooling mattress pad through comparing answers to subject questionnaires at baseline and follow up in addition to comparing the baseline diaries to the intervention diaries.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-60
* Peri or postmenopausal women (No periods for at least 3 months)
* Experiencing at least 4 hot flashes per day on average per week

Exclusion Criteria:

* Initiated CAM or non-CAM treatments for hot flashes in the last 4 weeks.
* Changed dose of a CAM or non-CAM treatments for hot flashes in the last 4 weeks
* Initiated antidepressants in the last 3 months.
* Changed their dose of an antidepressant in the last 3 months.
* Women who describe their health as fair or poor.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Avis, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Cooling Mattress Pad
Started | 38
Completed | 15
Not Completed | 23
Not completed — not eligbile after the 2-week diary | 9
Not completed — never returned their diary | 6
Not completed — dropped out of study before getting Chilipad | 5
Not completed — 3 did not complete follow-up questionnaire. | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population data includes only the participants who completed the study and who are included at baseline time frame in outcomes.
Arm/Group | Experimental Cooling Mattress Pad
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Diary
Description: Daily diary in which subjects will record the number of daily hot flashes and/or night sweats; reported as mean weekly number.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: number of hot flashes per week
Arm/Group | Experimental Cooling Mattress Pad
Number analyzed (Participants) | 15
number of hot flashes per week | 9 (4.5)

2. Primary Outcome: Hot Flash Diary
Description: as for outcome 1
Time Frame: Week 10
Population: 4 participants did not fill out hot flash diary at week 10
Measure: Mean (Standard Deviation); unit: number of hot flashes per week
Arm/Group | Experimental Cooling Mattress Pad
Number analyzed (Participants) | 11
number of hot flashes per week | 4.5 (3.0)

3. Primary Outcome: Hot Flash Severity Index Score
Description: The hot flash severity index score is a weighted total that combines number of hot flashes and severity using a 4- point severity scale from 1= mild to 4= very severe for each hot flash. Severity is calculated by multiplying the number of hot flashes by each level of severity. For example, 5 mild hot flashes would create a score of 5 and 3 very severe hot flashes would have a score of 12.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cooling Mattress Pad
Number analyzed (Participants) | 15
score on a scale | 20.0 (10.4)

4. Primary Outcome: Hot Flash Severity Index Score
Description: as for outcome 3
Time Frame: Week 10
Population: 4 did not fill out hot flash diaries at week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cooling Mattress Pad
Number analyzed (Participants) | 11
score on a scale | 7.8 (6.4)

5. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Questionnaire that assesses the subjects' quality of sleep through their answers to 19 questions on sleep quality. The global score ranges from 0 to 16 with a score >5 indicating poor sleep quality.
Time Frame: baseline
Population: 1 person did not answer all PSQI items at baseline, so data not included here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cooling Mattress Pad
Number analyzed (Participants) | 14
score on a scale | 11.14 (3.16)

6. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: as for outcome 5
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cooling Mattress Pad
Number analyzed (Participants) | 15
score on a scale | 7.87 (3.50)

7. Other Pre Specified Outcome: Hot Flash Related Daily Interference Scale (HFRDIS)
Description: Questionnaire that assesses interference that hot flashes cause in subjects' daily life. Scores range from 0-10 with a lower score being better.
Time Frame: baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Hot Flash Related Daily Interference Scale (HFRDIS)
Description: as for outcome 7
Time Frame: follow up at 11 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Center for Epidemiologic Studies Depression Scale (CESD-10)
Description: Questionnaire that assesses depression level (or lack of) in subjects. Scores range from 0-3 with a lower score being better.
Time Frame: baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Center for Epidemiologic Studies Depression Scale (CESD-10)
Description: as for outcome 9
Time Frame: follow up at 11 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Health Related Quality of Life (HRQL)
Description: Questionnaire that assesses quality of life in subjects. Score range 0-100 with a higher score being better.
Time Frame: baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Health Related Quality of Life (HRQL)
Description: Questionnaire that assesses quality of life in subjects. Score range 0-100 with a higher score being better.
Time Frame: follow up at 11 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Somatosensory Amplification Scale (SSAS)
Description: Questionnaire that assesses subject symptom sensitivity. Scores range 10-50 with a lower score being better.
Time Frame: baseline
Reporting Status: Not Posted

14. Other Pre Specified Outcome: General Anxiety Disorder (GAD-7)
Description: Anxiety symptoms will be measured with the GAD-7, which consists of 7 items, each describing a common symptom of anxiety. The respondent rates how much he or she has been bothered by each symptom over the past two weeks on a 4-point scale ranging from 0 to 3. Higher scores indicate more anxiety.
Time Frame: baseline and week 11
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Health Behaviors Questionnaire
Description: Questionnaire that allows the study team to record baseline behaviors
Time Frame: baseline
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Evaluation of Intervention
Description: Questionnaire that allows the study team to evaluate the subject's perception of how well the intervention worked.
Time Frame: follow up at 11 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline through week 10.
Arm/Group | Experimental Cooling Mattress Pad
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT03937466/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03937466/ICF_000.pdf